CLINICAL TRIAL: NCT02685618
Title: Safety and Efficacy of Low-dose Prostacyclin Administration and Blood Pressure Target in Addition to Standard Therapy, as Compared to Standard Therapy Alone, in Post-cardiac-arrest-syndrome Patients - a Randomized, Controlled, Double-blinded Investigator-initiated Trial.
Brief Title: Endothelial Dysfunction in Resuscitated Cardiac Arrest
Acronym: ENDO-RCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pär Johansson (Other)
Responsible Party: Sponsor-Investigator, Pär Johansson, MD, DMSc, MPA, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014092629
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Iloprost + M1006B offset by -10 mmHg (Experimental): Administration of 1 ng/kg/min Ilomedin® as a 48h continuous i.v infusion. Administration of blood pressure modules M1006B: offset by -10 mmHg
  Intervention: Drug: Iloprost + M1006B offset -10mmHg
  Interventions: Drug: Iloprost; Device: Phillips M1006B, offset by -10mmHg
- Iloprost + M1006B, No offset (Experimental): Administration of 1 ng/kg/min Ilomedin® as a 48h continuous i.v infusion Administration of blood pressure modules M1006B: No offset
  Intervention: Drug: Iloprost + M1006B, No offset
  Interventions: Drug: Iloprost; Device: Philips M1006B, No offset
- Placebo + M1006B offset by -10 mmHg (Placebo Comparator): Double dummy 0.9% saline as a 48h continuous i.v infusion. Administration of blood pressure modules M1006B: offset by -10 mmHg
  Intervention: Drug: Placebo + M1006B offset -10mmHg
  Interventions: Drug: Saline; Device: Phillips M1006B, offset by -10mmHg
- Placebo + M1006B, No offset (Placebo Comparator): Double dummy 0.9% saline as a 48h continuous i.v infusion Administration of blood pressure modules M1006B: No offset
  Intervention: Drug: Placebo + M1006B, No offset
  Interventions: Drug: Saline; Device: Philips M1006B, No offset

INTERVENTIONS:
Drug: Iloprost
  Other Names: Ilomedin (R); Prostacyclin analogue (PGI2)
  Arms: Iloprost + M1006B offset by -10 mmHg; Iloprost + M1006B, No offset
Drug: Saline
  Other Names: 0,9% NaCl
  Arms: Placebo + M1006B offset by -10 mmHg; Placebo + M1006B, No offset
Device: Phillips M1006B, offset by -10mmHg — Administration of blood pressure module M1006B: offset by -10 mmHg
  Arms: Iloprost + M1006B offset by -10 mmHg; Placebo + M1006B offset by -10 mmHg
Device: Philips M1006B, No offset — Administration of blood pressure module M1006B: No offset
  Arms: Iloprost + M1006B, No offset; Placebo + M1006B, No offset

SUMMARY:
Objective: Safety and efficacy of low-dose prostacyclin administration and blood pressure target in addition to standard therapy, as compared to standard therapy alone, in post-cardiac-arrest-syndrome (PCAS) patients.

DETAILED DESCRIPTION:
Trial Rationale: Therapeutic interventions directed towards the damaged endothelium may improve outcome for patients with PCAS. Prostacyclin/Iloprost (PGI2) is an endogenous prostanoid which is formed and released by endothelial cells with anti-platelet, vasodilatory and cytoprotective properties36 and is expected to be beneficial by protecting and deactivating the endothelium and by restoring vascular integrity in patients suffering from endothelial breakdown.

Trial Population: Participants in the trial must be adult patients (≥18 years of age) with out-of-hospital cardiac arrest (OHCA) of presumed cardiac cause admitted to the Dept. of Cardiology, 2143, Rigshospitalet, Copenhagen.

Trial Design: Randomized, placebo controlled, double-blind investigator-initiated trial in 40 OHCA patients. 48 hours of active study drug (Iloprost, 1 ng/kg/min) versus placebo (saline) infusion.

Patients in both randomization groups will be treated in accordance with state-of-the art therapy including targeted temperature management. Interventions are considered emergency procedures and study drug infusion should be commenced as soon as possible after sustained return of spontaneous circulation (ROSC), screening and randomization.

Patients will only be enrolled after informed consent, but as the treatment has to be initiated earliest possible after the out of hospital cardiac arrest diagnosis i.e., at a time-point where patients are temporarily incompetent, scientific guardians will co-sign the informed consent form before inclusion. Next-of-kin and the patients' general practitioner will co-sign as soon as possible and the patient will provide informed consent whenever possible.

During the study, blood samples will be taken at different time points. Patients will be observed and assessed continuously with regards to complications including bleeding. Patients will be actively assessed as long as the patient is in the ICU. During the extended follow up period at day 30, 90 and 180 contact will be made with the patients to follow up on safety events and vital status.

The trial is conducted in accordance with the protocol and is approved by Danish health and medicines authority, Danish ethics committee and danish data protection agency.

Investigational product: The active treatment in the trial is 1 ng/kg/min Ilomedin® administered as a 48h continuous i.v infusion. The drugs will be administered according to the product specifications.

Placebo: The placebo is 0.9% saline administered as a 48h continuous i.v infusion. The i.v volume of placebo saline to be administered is equal to the administered volume of diluted (in 0.9% saline) active drug.

Sponsor of study and financial support: This research project is investigator-initiated by the trial Sponsor Pär I. Johansson in collaboration with the principal investigator Christian Hassager.

It has not received funding from any commercial sponsors.

Patient recruitment period runs from February 2016 to August 2016. Follow-up data on 30-day, 90-day and 180-day outcome and adverse events will be collected. Initial data analyses will be done after completion of 30-day follow-up for all patients. Secondary data analyses will be done after completion of 180-day follow-up for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. OHCA of presumed cardiac cause
3. Sustained ROSC*
4. Unconsciousness (GCS <8) (patients not able to obey verbal commands) after sustained ROSC*
5. Target temperature management is indicated.

Exclusion Criteria:

1. Conscious patients (obeying verbal commands)
2. Females of childbearing potential (unless a negative human chorionic gonadotropin (HCG) test can rule out pregnancy within the inclusion window)
3. Patients weighing more than 135kg
4. In-hospital cardiac arrest (IHCA)
5. OHCA of presumed non-cardiac cause, e.g. after trauma or dissection/rupture of major artery OR Cardiac arrest caused by initial hypoxia (i.e. drowning, suffocation, hanging).
6. Known congenital bleeding diathesis (medically induced coagulopathy due to treatment with Vitamin K antagonists, Thrombininhibitors, Factor Xa inihbitors, ADP-receptor inhibitors, Aspirin, Asasantin, Persantin, NSAID, unfractionated and low molecular weight heparin does NOT exclude the patient).
7. Suspected or confirmed acute intracranial bleeding
8. Suspected or confirmed acute stroke
9. Unwitnessed asystole
10. Known limitations in therapy and Do Not Resuscitate-order
11. Known disease making 180 days survival unlikely
12. Known pre-arrest CPC 3 or 4
13. >4 hours (240 minutes) from ROSC to screening
14. Systolic blood pressure <80 mm Hg in spite of fluid loading/vasopressor and/or inotropic medication/intra-aortic balloon pump/axial flow device*
15. Temperature on admission <30°C.
16. Known allergy to Prostacyclin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Mean change i plasma biomarkers reflecting endothelial activation and damage | 48 hours
  Mean change in biomarkers indicative of endothelial activation and damage (sE-selectin, syndecan-1, soluble thrombomodulin (sTM), soluble vascular endothelial growth factor (sVEGF), nucleosomes) and sympathoadrenal overactivation (epinephrine/norepinephrine) from baseline to 48 hours post-randomization.

SECONDARY OUTCOMES:
Mean change in hemostatic profile evaluated by TEG, Multiplate, Flowcytometry | 48 hours
  Mean change in the hemostatic profile evaluated by Thrombelastography (TEG)(change in functional hemostatic blood test) and Multiplate (whole blood platelet aggregometry) and change in Flowcytometry (change in blood cell and endothelial cell derived microparticles). from baseline to 48 hours post-randomization.
Blood pressure target influence on primary outcomes measured by mean change in plasma biomarkers. | 48 hours
  Blood pressure target (65 mmHg or 75 mmHg) influence on the endothelial response to the study drug (mean change in biomarkers reflecting endothelial activation and damage) and change in levels of Neuron Specific Enolasis from baseline to 48 hours post-randomization.
Feasibility of blood pressure target intervention. | 48 hours
  Feasibility of blood pressure target intervention .(Target 90%)

OTHER OUTCOMES:
Number of patients with severe bleeding | 24 hours-180 days
  Severe bleeding (intracranial or clinical bleeding with the use of 3 red blood cells (RBC) units or more/24 hours)
Number of patients requiring organ support | 48 hours to 180 days
  Days of vasopressor, ventilator and renal replacement therapy post-randomization.
Mean change in disease severity score | 48 to 96 hours
  Changes in SOFA score from baseline to 48 h and day 4 post-randomization.
Number of patients with transfusion requirements | 48 hours to 180 days
  Use of blood products (in ICU) post-randomization.
Grading of Neurological function. | to 180 days
  Neurological function graded by modified Rankin Scale (mRS) and Cerebral Performance Category (CPC) at 180 days.
Mortality | 24 hours to 180 days
  Difference in day 7, 30, 90 and 180 day mortality between patients receiving active treatment (lloprost) and placebo.
Evaluation of Renal function | 24 to 96hours
  Estimated glomerular filtration rate (eGFR) and urine output at day 2 and 3 and need for renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chistian Hassager, MD, DMSc, Principal Investigator — Dept. of Cardiology, 2143, Rigshospitalet, Blegdamsvej 0, DK-2100
Locations (1):
- Dept. of Cardiology, 2143, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Meyer ASP, Ostrowski SR, Kjaergaard J, Frydland M, Thomsen JH, Johansson PI, Hassager C. Low dose Iloprost effect on platelet aggregation in comatose out-of-hospital cardiac arrest patients: A predefined sub-study of the ENDO-RCA randomized -phase 2- trial. J Crit Care. 2020 Apr;56:197-202. doi: 10.1016/j.jcrc.2019.12.025. Epub 2019 Dec 30. PMID 31945586
- [Derived] Meyer ASP, Johansson PI, Kjaergaard J, Frydland M, Meyer MAS, Henriksen HH, Thomsen JH, Wiberg SC, Hassager C, Ostrowski SR. "Endothelial Dysfunction in Resuscitated Cardiac Arrest (ENDO-RCA): Safety and efficacy of low-dose Iloprost, a prostacyclin analogue, in addition to standard therapy, as compared to standard therapy alone, in post-cardiac-arrest-syndrome patients.". Am Heart J. 2020 Jan;219:9-20. doi: 10.1016/j.ahj.2019.10.002. Epub 2019 Oct 21. PMID 31710844
- [Derived] Meyer AS, Ostrowski SR, Kjaergaard J, Johansson PI, Hassager C. Endothelial Dysfunction in Resuscitated Cardiac Arrest (ENDO-RCA): safety and efficacy of low-dose prostacyclin administration and blood pressure target in addition to standard therapy, as compared to standard therapy alone, in post-cardiac arrest syndrome patients: study protocol for a randomized controlled trial. Trials. 2016 Aug 2;17:378. doi: 10.1186/s13063-016-1477-z. PMID 27484224